CLINICAL TRIAL: NCT02799979
Title: 3D Imaging: Prognostic Role in Pulmonary Arterial Hypertension
Acronym: HTP3S
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Other Study IDs: 14-AOI-08
Record Dates: First submitted 2016-05-30; First posted 2016-06-15 (Estimated); Last update posted 2017-10-05 (Actual); Status verified 2017-10

CONDITIONS: Pulmonary Arterial Hypertension
MeSH Terms: conditions — Pulmonary Arterial Hypertension

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Case: Echocardiographic data : 3D right ventricular imaging on 100 pulmonary hypertension patients at Baseline and after six months
  Interventions: Device: 3D right ventricular imaging echocardiographic
- Control: Echocardiographic data : 3D right ventricular Imaging on 50 patients without pulmonary hypertension only at baseline
  Interventions: Device: 3D right ventricular imaging echocardiographic

INTERVENTIONS:
Device: 3D right ventricular imaging echocardiographic — Echocardiographic data (3D right ventricular imaging echocardiographic) will be collected at baseline and after 6months.

SUMMARY:
Pulmonary hypertension is a rare and severe disease, affecting a young population. Survival is very poor and has been closely related to right ventricular dysfunction. Current prognostic equations rely mostly on right heart catheterization data. The identification of simple echocardiographic prognostic factor is urgently needed. It could help identifying with a non invasive method, high risk patients who could benefit from an intensive specific therapy. 3D right ventricular imaging is a new echocardiographic tool which provides RV volumic analysis, RV ejection fraction, overcoming the classical limits of 2D ultrasound.

The aim of this study is to validate a new software for 3D analysis of the right ventricle and assess its prognostic role in pulmonary hypertension.

To do so, the investigators will realize a prospective monocentric longitudinal cohort study, including 100 pulmonary hypertension patients. Echocardiographic data will be collected at baseline and after 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients > 18 years old
* Pulmonary hypertension diagnosed by right heart catheterization
* Informed consent obtained
* Affiliation to the French national health insurance

Exclusion Criteria:

* Associated significant left heart disease
* Sub-optimal acoustic windows
* Patient unable to attend follow-up visits

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with pulmonary hypertension diagnosed
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2014-10; Primary Completion 2018-10 (Estimated); Study Completion 2019-06 (Estimated)

PRIMARY OUTCOMES:
Number of death from any cause | Baseline to 24 months
  Description of the number of death during the study

SECONDARY OUTCOMES:
Number of Hospitalisation | Baseline to 24 months
  Description of the number of hospitalisation for worsening of pulmonary arterial hypertension
3D right ventricular imaging echocardiographic | Baseline and 6 months
  Analyse the data of 3D right ventricular (RV), ejection fraction, RV telediastolic and telesystolic volume, 3D RV area strain (%)

CONTACTS AND LOCATIONS:
Overall Officials: PAMELA MOCERI, MD, Principal Investigator — CHU NICE
Locations (1):
- Hopital Pasteur - Chu Nice, Nice, France

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Moceri P, Duchateau N, Baudouy D, Squara F, Bun SS, Ferrari E, Sermesant M. Additional prognostic value of echocardiographic follow-up in pulmonary hypertension-role of 3D right ventricular area strain. Eur Heart J Cardiovasc Imaging. 2022 Oct 20;23(11):1562-1572. doi: 10.1093/ehjci/jeab240. PMID 36265185